CLINICAL TRIAL: NCT06570473
Title: Feasibility Trial for the Canadian Right Ventricular AdaptiVE (CRAVE) Platform for Therapies Targeting Right Ventricular Failure
Brief Title: Feasibility Trial for a Right Ventricular Failure Platform Trial
Acronym: CRAVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Heart Function Alliance (Unknown); Accelerating Clinical Trials Consortium (Other); Ottawa Heart Institute Research Corporation (Other); Team PHenomenal Hope (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAVE-01
Record Dates: First submitted 2024-08-21; First posted 2024-08-26 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Hypertension; Right Ventricular Dysfunction; Right Heart Failure
Keywords: Pulmonary Hypertension; Right Ventricular Dysfunction; Right Heart Failure; Empagliflozin; Ranolazine
MeSH Terms: conditions — Hypertension, Pulmonary; Ventricular Dysfunction, Right; Heart Failure | interventions — empagliflozin; Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Empagliflozin (Experimental): Participants in the empagliflozin arm will receive 10 mg by mouth once daily and standard of care.
  Interventions: Drug: Empagliflozin
- Ranolazine (Experimental): Participants in the ranolazine arm will receive ranolazine 500 mg by mouth twice daily, which will be increased to 1000 mg twice daily after 2 weeks (unless concurrently using moderate CYP 3A4 inhibitors, then dose is limited to 500 mg twice daily) and will receive standard of care.
  Interventions: Drug: Ranolazine
- Standard of Care (No Intervention): Participants in this group will receive standard of care.

INTERVENTIONS:
Drug: Empagliflozin — Tablet
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Ranolazine — Tablet
  Other Names: Corzyna
  Arms: Ranolazine

SUMMARY:
The primary objective of the CRAVE feasibility trial is to assess the feasibility of conducting a larger CRAVE platform trial by performing a randomized trial of 30 participants with pulmonary hypertension and right ventricular dysfunction, comparing empagliflozin or ranolazine plus standard of care to standard of care alone.

DETAILED DESCRIPTION:
This study is an investigator-initiated, open label, prospective, multi-centre, phase 2, randomized control trial. This CRAVE feasibility trial will seek to establish the feasibility of a larger platform trial for testing multiple interventions in various domains to improve right ventricular function. In this feasibility trial, 30 participants with pulmonary hypertension and right heart failure with be randomized 1:1:1 to empagliflozin 10 mg daily + standard of care, ranolazine twice daily + standard of care, or standard of care alone. Participant outcomes (medical records review) will be followed for 16 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to provide informed consent.
3. Able to comply with all study procedures.
4. History of RV dysfunction or RHF secondary to any of:

   a. Group 1 PH, pulmonary arterial hypertension b. Group 2 PH, left heart disease with normal left ventricular ejection fraction (LVEF) > 50% and a previous RHC demonstrating combined pre and post-capillary PH, defined as: i. mPAP >20 mmHg ii. PAWP > 15 mmHg iii. PVR> 2 WU c. Group 3 PH d. Group 4 PH, chronic thromboembolic PH that is either persistent after pulmonary endarterectomy or inoperable due to distal disease.
5. Symptomatic with current NYHA Functional Class II-IV
6. Biomarker and 2D echocardiogram evidence of RV dysfunction within 3 months:

   1. NT-proBNP >300 ng/L and qualitative evidence of at least 'mild' RV dysfunction on echocardiography OR NT-proBNP<300 ng/L and qualitative evidence of at least moderate RV dysfunction and/or dilatation on 2D echocardiogram AND
   2. A quantitative 2D echocardiogram with evidence of RV dysfunction defined as having both of the following:

   i. TAPSE ≤18 mm ii. RV dilatation (RV diameter > 42 mm at the base).
7. Receiving loop diuretics or mineralocorticoid receptor antagonists for at least 4 weeks.
8. Access to an iOS or android smart phone or tablet.

Exclusion Criteria:

1. Estimated glomerular filtration rate (eGFR) <30 ml/min.
2. LVEF < 50%
3. Normal RV size and function
4. Severe aortic or mitral valvular disease
5. Moderate or severe hepatic dysfunction (Child-Pugh Class B or C)
6. Participants requiring augmentation of diuretics or otherwise not meeting definition for clinical stability
7. Pregnancy or lactation
8. Unable to provide consent and comply with follow-up visits
9. Listed for lung, heart or heart/lung transplantation
10. Myocardial infarction or acute coronary syndrome within 90 days of screening
11. Enrolled in another interventional trial
12. Planned cardiac or thoracic surgical intervention in the next 6 months.
13. Known hypersensitivity to empagliflozin or ranolazine.
14. Concurrent treatment with:

    * strong inhibitors of Cytochrome P450 3A4 (CYP 3A4), (e.g., ketoconazole, itraconazole, voriconazole, posaconazole, clarithromycin, nelfinavir, ritonavir, indinavir, saquinavir and grapefruit juice)
    * class IA antiarrhythmics (e.g., quinidine, procainamide, disopyramide) or class III antiarrhythmics (e.g., sotalol, ibutilide, amiodarone, dronedarone)
    * inducers of CYP 3A4 (e.g., rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine, and St. John's wort)
15. Congenital long QT syndrome or a QTc interval >500 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of eligible participants approached that consent | 16 weeks
  (target ≥30%)
The proportion of participants who consent that are randomized | 16 weeks
  (target ≥90%)
Average enrolment rate of participants per centre per month | 16 weeks
  (target ≥1 participant per centre/month)
Loss of follow up or death | 16 weeks
  Loss of follow up (target at 16 weeks ≤5%)
Ability to capture data for secondary outcomes | 16 weeks
  (target ≥90% completion)

SECONDARY OUTCOMES:
RV function | 16 weeks
  assessed using echocardiogram
Natriuretic peptides | 16 weeks
  (N-terminal pro-B-type natriuretic peptide [NT-proBNP])
Hemodynamics | 16 weeks
  assessed using right heart catheterization (RHC)
Exercise capacity measured virtually | 16 weeks
  6-minute walk distance (6MWD) assessed using the novel Walk.Talk.Track. mobile app
Exercise capacity measured in-person | 16 weeks
  assessed using in-person 6-minute walk distance (6MWD)
NYHA functional class | 16 weeks
  (New York Heart Association Functional Classification for heart failure)
EmPHasis-10 | 16 weeks
  questionnaire used during clinical assessments to determine how pulmonary hypertension affects someone's life
KCCQ-12 | 16 weeks
  questionnaire for assessing health-related quality of life in chronic heart failure
EQ-5D-5L | 16 weeks
  questionnaire provides a simple descriptive profile of a respondent's health state
Clinical event outcomes | 16 weeks
  number of clinical events that occur

CONTACTS AND LOCATIONS:
Overall Officials: Jason Weatherald, MD,MSc,FRCPC, Principal Investigator — University of Alberta
Locations (5):
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - The University of British Columbia, Vancouver, British Columbia
  - London Health Sciences Centre - University Hospital, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.